CLINICAL TRIAL: NCT06474195
Title: Effectiveness of Cue-based Intervention in Improving Prospective Memory by Enhancing Medication Adherence in Patients With Schizophrenia and Schizoaffective Disorder: A Randomized Controlled Trial
Brief Title: Cue-based Intervention in Prospective Memory and Medication Adherence.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); St.John's Medical College and Hospital (Unknown)
Responsible Party: Principal Investigator, Vishwajit Nimgaonkar, MD PhD, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY22120098; D43TW009114 (NIH)
Record Dates: First submitted 2024-06-18; First posted 2024-06-25 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Schizophrenia
Keywords: Adherence; Schizophrenia; Cue based
MeSH Terms: conditions — Schizophrenia | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled study. The participants will be randomly assigned to treatment as usual arm or intervention arm. The intervention arm will receive the cues in the form of daily repeating reminders for a time period of 30 days. The participant will also be asked a task of daily routine during the same time of medication. The Treatment as Usual (TAU) Arm will not get any reminders but the baseline assessment will be similar to the intervention arm. There will be 2 follow-ups, 1st follow-up will be 30 days after the baseline assessment and the second will be 90 days after the baseline assessment. repeated during both follow-up visits. TAU will also be followed up at 30 days and 90 days after baseline assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): . The intervention arm will receive the cues in the form of daily repeating reminders for a time period of 30 days. The reminders will be set on participants' mobile phones to receive at least 1 hour prior to the prescribed oral antipsychotic medication. The same reminder will be repeated after 10 minutes duration to ensure that the participant does not miss the cue and the uniformity of the cue will be ensured by setting the same emoji or the same phrase on the participant's own mobile phone. The participant will also be asked a task of daily routine during the same time of medication.
  Interventions: Behavioral: Cue based intervention
- Treatment as Usual (Active Comparator): Treatment as Usual (TAU) Arm will not get any reminders but the baseline assessment will be similar to the intervention arm.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Cue based intervention — The intervention arm will receive the cues in the form of daily repeating reminders for a time period of 30 days. The reminders will be set on participants' mobile phones to receive at least 1 hour prior to the prescribed oral antipsychotic medication. The same reminder will be repeated after 10 minutes duration to ensure that the participant does not miss the cue and the uniformity of the cue will be ensured by setting the same emoji or the same phrase on the participant's own mobile phone. The participant will also be asked a task of daily routine during the same time of medication.
  Arms: Intervention
Behavioral: Treatment as Usual — This group will not get any intervention but the usual treatment all assessments will continue
  Other Names: TAU
  Arms: Treatment as Usual

SUMMARY:
Medication adherence is a major challenge while treating patients with major mental illnesses like schizophrenia and schizoaffective disorder. This interventional study aims to assess the improvement in prospective memory and thus medication adherence by giving time and event-based cues to the participants.

DETAILED DESCRIPTION:
According to available evidence, prospective memory (PM) is important in daily functioning but is impaired in schizophrenia. However, there were hardly any Indian studies on this topic. Medication adherence is one of the challenges which clinicians often face during treatment. Our study aims to enhance medication adherence and prospective memory using a cue-based intervention.

Aims:

To assess the improvement in prospective memory using cue-based intervention to enhance medication adherence and basic functional skills.

Objective:

1. To correlate prospective memory and medication adherence with executive function and cognitive insight.
2. To correlate the medication adherence with basic functional skills

Hypotheses to be tested:

1. Statistically significant difference between prospective memory improvement with intervention in the intervention group and treatment as usual group.
2. A Statistically significant correlation between prospective memory score and medication adherence score.
3. A Statistically significant correlation between medication adherence and basic functional skills.

The study will have two arms with two arms (n=52 in each group) the intervention arm and the TAU arm. Participants in both arms will receive standard medical care as advised by the treating psychiatrist. The treating psychiatrist will be blinded about which group the patient belongs to and they will be encouraged to prescribe stable medication throughout the study process unless it would affect the treatment outcome or prognosis of the patient. The intervention arm will receive the cues in the form of daily repeating reminders for a time period of 30 days. The reminders will be set on participants' mobile phone to receive at least 1 hour prior to the prescribed oral antipsychotic medication. The same reminder will be repeated after 10minutes duration to ensure that participant does not miss the cue and the uniformity of the cue will be ensured by setting the same emoji or the same phrase on the participants own mobile phone. The participants will also be encouraged to close their eyes for 5-7 seconds and imagine themselves to be taking the medication at the prescribed time when they see the reminder. The family members or the caretaker of the patient will be provided with a adherence chart which will be reviewed during the follow up visits. During the baseline assessment Independent Living Skills Survey (ILSS) questionnaire will be administered to obtain a baseline score of living skills and the domain with least score will be addressed by individual based intervention using similar cue-based intervention by repeated reminders will be done to improve that domain and during the follow up visit the improvement will be assessed by comparing the follow up scores of (ILSS) with baseline scores. Subsequently on first follow up the medication adherence will be assessed using Brief Adherence Rating Scale (BARS) and prospective memory will be assessed using Memory for Intentions Screening Test (MIST) and the score will be briefed to the patients and patients will be motivated to comply with study process till the second follow up. The second follow up assessment will be done after 90 days from baseline assessment. During the time period between first and second follow up the participants will not receive any cue. Participants will be assessed using Memory for Intentions Screening Test (MIST), Brief Adherence Rating Scale (BARS), Trail Making Test (TMT), Beck Cognitive Insight Scale (BCIS) and Independent Living Skills Survey (ILSS) during baseline, first follow up and second follow up. During each sessions patients as well as family will be enquired if they suffered from any distress related to the study, both psychological and physical. In that case it will be explored in detail and if required necessary intervention will be given after after consulting with the treating psychiatrists.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female age 18 - 60 years

  * Diagnosed with Schizophrenia as per DSM V Criteria
  * Insight of grade 3 or more.
  * At least 10th standard level of education in the English language

Exclusion Criteria:

* Comorbid chronic medical illnesses.
* Psychoactive substance use in harmful use pattern or in dependence pattern.
* Co-existing neurodevelopmental disorders or learning disorders.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Prospective memory | Baseline, After 30days' intervention
  Change in prospective memory in intervention arm as measured by compared to TAU The Memory for Intentions Screening Test(MIST) score as compared to TAU
Prospective memory (sustainability) | Baseline, 90 days after baseline assessment
  Change in prospective memory in intervention arm as measured by compared to TAU The Memory for Intentions Screening Test (MIST) score as compared to TAU
Medication adherence | Baseline, After 30days' intervention
  Change in medication adherence in intervention arm as measured by Brief Adherence Rating Scale (BARS) score as compared to TAU
Medication adherence (Sustainability) | Baseline, 90 days after baseline assessment
  Change in medication adherence in intervention arm as measured by Brief Adherence Rating Scale (BARS) score as compared to TAU

SECONDARY OUTCOMES:
Cognition | Baseline, After 30days' intervention
  Change in cognition in intervention arm as measured by Trail Making Test (TMT) score as compared to TAU
Cognition (Sustainability) | Baseline, 90 days after baseline assessment
  Change in cognition in intervention arm as measured by Trail Making Test (TMT) score as compared to TAU
Independent living skills score | Baseline, After 30days' intervention
  Change in Independent living skills score in intervention arm as measured by Independent living skills scale (ILSS) score as compared to TAU
Independent living skills score (Sustainability) | Baseline, 90 days after baseline assessment
  Change in Independent living skills score in intervention arm as measured by Independent living skills scale (ILSS) score as compared to TAU
Cognitive Insight | Baseline, After 30days' intervention
  Change in Independent living skills score in intervention arm as measured by Cognitive Insight Scale (BCIS) score as compared to TAU
Cognitive Insight (Sustainabilty) | Baseline,90 days after baseline assessment
  Change in Independent living skills score in intervention arm as measured by Cognitive Insight Scale (BCIS) score as compared to TAU

CONTACTS AND LOCATIONS:
Overall Officials: Vishwajit L Nimgaonkar, MD, PhD, Principal Investigator — University of Pittburgh
Locations (1):
- St. John's Medical College and Hospital, Bengaluru, Karnataka, India

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: One year after publication of this study.
Access Criteria: For individual participant data, meta-analysis.